CLINICAL TRIAL: NCT07199634
Title: Integrating U=U Into HIV Counseling in South Africa (INTUIT-2.0): a Cluster-Randomized Trial
Brief Title: Integrating U=U Into HIV Counseling in South Africa (INTUIT-2.0)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H-46247; 1R01MH135774-01A1 (NIH)
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: HIV
Keywords: HIV Counseling South Africa; Antiretroviral treatment (ART); Person living with HIV (PLWH); Undetectable=Untransmittable (U=U); Viral load

STUDY DESIGN:
Intervention Model Description: The study will be a cluster-randomized trial (CRT), where clinics are pair-matched and randomized into immediate intervention (Group A) and deferred intervention (Group B, control) groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate intervention Group A (Experimental): Participants whose clinic was randomized into Group A will have immediate access to the "Undetectable & You" intervention app as part of HIV counseling.
  Interventions: Other: "Undetectable & You" HIV treatment literacy app
- Deferred intervention Group B (Active Comparator): Participants whose clinic was randomized into Group B will get the intervention app at 16 months, after data collection for primary outcomes is complete.
  Interventions: Other: "Undetectable & You" HIV treatment literacy app

INTERVENTIONS:
Other: "Undetectable & You" HIV treatment literacy app — The app delivers information on the transmission prevention benefits of HIV treatment through the Undetectable Equals Untransmutable (U=U) message, alongside real-life video testimonials of patients living with HIV (PLHIV) and their partners. It underscores the key behavioral skills required for U=U, namely, ART adherence and viral load monitoring.

SUMMARY:
Undetectable = Untransmittable (U=U) is the scientific consensus that people with human immunodeficiency virus (HIV) who achieve viral suppression through antiretroviral treatment (ART) cannot transmit the virus sexually. While global studies confirm this, awareness of U=U remains very limited in sub-Saharan Africa, including South Africa, where only two-thirds of people living with HIV (PLHIV) are virally suppressed despite having the largest treatment program globally. Many PLHIV delay or avoid ART because they feel healthy and perceive little benefit, while also fearing stigma, disclosure, and social costs. U=U offers powerful motivation for ART uptake and adherence by reframing treatment as both a personal health and prevention tool, reducing internalised stigma, strengthening self-image, and supporting HIV prevention altruism. Yet, dissemination in Africa has lagged. To address this, the investigators developed an HIV treatment literacy App called "Undetectable & You", which delivers accurate U=U information alongside real-life video testimonials of PLHIV and their partners. This research will assess the impact of the "Undetectable & You" App in a cluster-randomized trial in South Africa. The study will establish whether disseminating U=U information via a video-based app at the time of HIV counselling improves retention in care and viral suppression among PLHIV in South Africa.

Aim 1. Refine the "Undetectable & You" App to help PLHIV navigate U=U within relationships.

Aim 2. Establish the real-world impact of "Undetectable & You" on retention on ART and viral suppression in a cluster-randomized trial.

DETAILED DESCRIPTION:
The study will be a cluster-randomized trial (CRT), where clinics are pair-matched and randomized into immediate intervention (Group A) and deferred intervention (Group B, control) groups. The rationale for this design is to assess the impact of the Undetectable & You app-based HIV counselling intervention while ensuring that all clinics eventually receive the intervention. The deferred intervention control condition ensures that comparison clinics continue providing standard-of-care HIV counselling during the initial phase of the trial, without exposure to the Undetectable & You app. This allows for a comparison between the intervention and control groups while controlling for external factors.

Data will be collected from an Active Recruitment Cohort (ARC) (n=880) including survey data linked to routine clinical and laboratory records. The primary outcome is documented HIV viral load <200 copies/mL at 3-9 months after entry into the study. Secondary outcomes include documented HIV viral load <200 copies/mL at 9-15 months, any viral monitoring at 3-9months and 9-15months, and retention in care (any medication pick-ups) at 5-6 months and at 11-12 months. In addition to the ARC, a Passive Surveillance Platform (PSP) using de-identified South African National Health Laboratory Service (NHLS) data (N ~28,000) will allow for higher-powered assessment of impacts on viral suppression across all patients at study clinics.

ELIGIBILITY:
Inclusion Criteria-

Clinic inclusion criteria:

* Public sector facility
* Primary care, outpatient clinic
* Follows national guidelines for HIV counseling
* Has dedicated HIV counselors
* At least 10 patients receiving HIV counseling per week (based on pre-study data)
* Follows national guidelines for lab monitoring (CD4 at diagnosis; VLs at 3 and 10 months on ART)
* Is interested in participating, as indicated by "sign-off" from the head nurse / facility director

Individual participant inclusion criteria:

* Adult (at least 18 years)
* Received HIV post-test counselling or adherence counseling
* Able to consent
* Provides informed consent
* Speaks one of the primary study languages: English, Zulu, Sotho, Tsonga
* Receives care at the facility as evidence by having a clinical record there

Individual participant exclusion Criteria:

* Require acute medical care that would be hindered by participation in the study
* Determined by clinical staff not to be physically or emotionally able to initiate ART
* Children (under 18 years).
* Prisoners or other institutionalized persons.
* Do not speak one of the primary study languages: English, Zulu, Sotho
* Are not able to consent (e.g. intoxicated or of limited mental capacity)
* Do not consent to participate in the study, including linkage to clinical records for follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 880 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2028-04-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
HIV viral load <200 copies/mL | 3-9 months (on average 6 months)
  Abstracted from clinical and laboratory records.

SECONDARY OUTCOMES:
HIV viral load <200 copies/mL | 9-15 months (on average 12 months)
  Abstracted from clinical and laboratory records.
Any viral monitoring | 3-9 months (on average 6 months), 9-15 months (on average 12 months)
  Abstracted from clinical and laboratory records.
Retention in care | 5-6 months, 11-12 months
  Retention in care is defined as any medication pick-ups by participants and will be abstracted from the clinical records.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Bor, Principal Investigator — BU School of Public Health, Global Health; Dorina Onoya, PhD, MBA, Principal Investigator — University of Witwatersrand, South Africa

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD will be posted to a public repository, e.g. OSF.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: IPD and supporting information will be posted when our primary outcomes paper is published.
Access Criteria: IPD and supporting information will be accessible to the public.